CLINICAL TRIAL: NCT03481699
Title: Prevention of Depression and Bullying in Adolescents by Means of an Intervention Based on Implicit Theories of Personality
Brief Title: Intervention Based on Implicit Theories of Personality: Effects on Depression and Bullying
Acronym: ITP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Deusto (Other)
Collaborators: Medikosta IMQ Análisis Clínicos (Unknown)
Responsible Party: Principal Investigator, Esther Calvete, Principal Investigator, Deusto Stress Research Team, University of Deusto, University of Deusto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PSI2015-68426-R
Record Dates: First submitted 2018-03-20; First posted 2018-03-29 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Depression; Bullying
Keywords: Adolescence; Prevention; Emotional disorders; Aggressive behavior
MeSH Terms: conditions — Depression; Bullying; Aggression | interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: Participants were randomized in a 1:1 ratio blocked by gender to one of two groups: experimental condition (ITP intervention) versus control condition (educational intervention) in parallel for the duration of the study.
Who Masked: Participant, Outcomes Assessor
Masking Description: Allocation was concealed to the participants, researchers -who were in class the assessment days- and teachers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Incremental theory of personality (Experimental): 1 hour behavioral intervention (based on ITP) consisting on several tasks to be completed on paper individually.
  Interventions: Behavioral: Incremental theory of personality
- Educational intervention (Other): 1 hour educational intervention (about the human brain) consisting on several tasks to be completed on paper individually.
  Interventions: Other: Educational Intervention

INTERVENTIONS:
Behavioral: Incremental theory of personality — The experimental intervention (originally developed by David S. Yeager and colleagues) teaches that individuals have the potential to change. It has three main parts. First, participants are asked to read scientific studies that provide evidence that behaviors are controlled by "thoughts and feelings in brains," and that pathways in the brain have the potential to be changed under the right circumstances. Second, participants read several testimonials purportedly written by upperclassmen to bring credibility to the ITP. Finally, participants are asked to write their own version of such a narrative. This self-persuasive writing exercise has been shown to facilitate the internalization of the intervention message, building on a long line of research on cognitive dissonance.
  Arms: Incremental theory of personality
Other: Educational Intervention — The educational intervention involved scientific information about the human brain. It was designed to be parallel to the experimental intervention and, hence, it has also three main parts. First, participants are asked to read scientific information about the different areas of the brain and their specialties. Second, participants read several testimonials written by upperclassmen about their transition to high school and how their brains help them to adapt to the new space and all the physical differences of the building and the classes. Finally, participants are asked to write a letter to another student explaining the main things he or she has learned about the brain and thinks are important for adapting to the new physical environment in high school.
  Arms: Educational intervention

SUMMARY:
This study evaluates the efficacy of an intervention based on the Implicit Theories of Personality (ITP) in Spanish adolescents. Half of participants received the ITP intervention, while the other half received an educational intervention.

DETAILED DESCRIPTION:
Depression and bullying are two problems arising in childhood and adolescence, which cause severe suffering. Although there are good intervention programs for children and adolescents at risk, the results for universal interventions have generally been poor. The current project will test the efficacy of an Intervention based on the Implicit Theories of Personality (ITP). This procedure has recently been developed at US by David S. Yeager and colleagues, with extraordinary results in the reduction of depression, stress, and aggression. The project includes the following aims: (1) the evaluation of the efficacy of the ITP on depressive symptoms (Study 1) and aggressive behavior (Study 2) in Spanish adolescents; (2) to test whether the intervention changes biological and cognitive variables; (3) to identify whether development and sex moderates the effects of the intervention; and (4) to test whether temperament moderates the effect of the intervention. The study involves the evaluation of the intervention in a sample of around 900 adolescents (12-18 years), randomly allocated to experimental and control condition. It is a field experiment conducted in high schools and involves multiple measures over time (self-reports and parent reports; as well as levels of cortisol, testosterone and DHEA in saliva in a subset -50%- of the participants). In summary, the project aims to respond to the challenge of health and wellness in the population through a randomized controlled trial with multiple sources of measure and from a biopsychosocial perspective. The ITP intervention has the potential to become a universal intervention to help reduce the rates of depression and bullying.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent by the adolescents and their parents.
* To be fluent in Spanish.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 882 (Actual)
Dates: Start 2016-10-03 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline scores of the Center for Epidemiologic Studies Depression scale (CES-D; Radloff, 1977) at 2 weeks, 6 months, and 12 months. | Baseline, 2 weeks, 6 months, and 12 months.
  Self reported depressive symptoms during the last month (last week in the 1 week follow-up) measured by 20 items scored 0-3 (0 = rarely; 3 = most or almost all the time), yielding a total between 0 and 60.
Change from baseline scores of the Revised version of the Peer Experiences Questionnaire (RPEQ; Prinstein, Boergers, & Vernberg, 2001) at 2 weeks, 6 months, and 12 months. | Baseline, 2 weeks, 6 months, and 12 months.
  Self reported levels of perpetration (9 items) of peer aggression in the school context during the last 6 months (last week in the 1 week follow-up). Each item is scored 1-5 (1 = never; 5 = several times per week), yielding a total between 18 and 90.
Change from baseline scores of the Cyber Bullying Questionnaire (CBQ; Calvete et al., 2012; Gámez-Guadix, Villa-George, & Calvete, 2014) at 2 weeks, 6 months, and 12 months. | Baseline, 2 weeks, 6 months, and 12 months.
  Self reported levels of perpetration (9 items) of peer cyber aggression during the last 6 months (last week in the 1 week follow-up). Each item is scored 0-3 (0 = never; 3 = five or more times), yielding a total between 0 and 54.
Change from baseline levels of Cortisol, DHEA and testosterone (in saliva) at 2 weeks, 6 months, and 12 months. | Baseline, 2 weeks, 6 months, and 12 months.
  A random subset of the participants (n = 546) have provided saliva samples to be assayed for neuroendocrine levels to measure cortisol, DHEA and testosterone. They were directed to transfer saliva from their mouths to a tube. The sample tubes were carefully labelled, and as soon as the session ended, saliva samples were sent to the assay laboratory (Medikosta IMQ Análisis Clínicos) and stored in a freezer at -80°C.

OTHER OUTCOMES:
Implicit Theories of Personality questionnaire (Yeager et al., 2014) | Baseline, 2 weeks, 6 months, and 12 months.
  Self reported measure that assesses adolescents' implicit theories of personality during the last 6 months (last week in the 1 week follow-up) measured by 8 items scored 1-6 (1 = strongly disagree; 6 = strongly agree), yielding a total between 8 and 48.
Young Schema Questionnaire (YSQ-3; Young, 2006) | Baseline, 2 weeks, 6 months, and 12 months.
  Self reported maladaptive cognitive schemas during the last 6 months (last week in the 1 week follow-up). The original version has 90 items, but for the purposes of this study, we have included 35 items of 7 subscales: defectiveness/shame (5 items), mistrust/abuse (5 items), entitlement superiority/grandiosity (5 items), failure to achieve (5 items), insufficient self control/self discipline (5 items), abandonment/instability (5 items), emotional deprivation (deprivación). Each item is scored 1-6 (1 = strongly disagree; 6 = strongly agree), yielding a total between 5 and 30 for each subscale.
Big Five Questionnaire for children (BFQ-C; Barbaranelli et al., 2003) | Baseline.
  Self reported questionnaire that assesses five personality traits: openness to experience, conscientiousness, extraversion, agreeableness, and neuroticism. For the purpose of this study, we have used the 21 items from the extraversion and neuroticism subscales. Each item is scored 1-5 (1 =almost always untrue of you ; 5 = almost always true of you).
Revised version of the Early Adolescent Temperament Questionnaire (EATQ-R; Ellis and Rothbart, 2001). | Baseline.
  Self reported questionnaire of that assesses temperament in adolescents. For this study, only the 10 items of the temperament domain of effortful control were used, which measure self-regulation aspects of temperament in adolescents with three subscales: inhibition control, attention and activation control. Each item is scored 1-5 (1 =almost always untrue of you ; 5 = almost always true of you), yielding a total between 1 and 50.

CONTACTS AND LOCATIONS:
Overall Officials: Esther Calvete, PhD, Principal Investigator — University of Deusto

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will be provided to the journals in which it is planned to publish the results of the study. In addition, the PI and research team will consider to make IPD available to other researchers after publishing the results of the study.

DOCUMENTS (2):
  • Informed Consent Form (2016-09-01): https://cdn.clinicaltrials.gov/large-docs/99/NCT03481699/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2016-09-01): https://cdn.clinicaltrials.gov/large-docs/99/NCT03481699/Prot_SAP_003.pdf